CLINICAL TRIAL: NCT00383110
Title: Racial/Ethnic Differences in Trust/Mistrust and Its Effect on Diabetes Outcomes
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: LIP 82-001; HR#11259 (Other: MUSC/VA IRB)
Record Dates: First submitted 2006-09-28; First posted 2006-10-02 (Estimated); Results first posted 2014-09-17 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2014-06

CONDITIONS: Diabetes
Keywords: Diabetes; Health Outcomes; Racial Preference; Clinical Trial; Ethnic Differences
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Adults (age 18 or older) with type 2 diabetes.

SUMMARY:
1. Determine racial/ethnic differences in trust in physicians and mistrust of the health care system among veterans with Type 2 Diabetes.
2. Determine the predictive power of trust in physicians and mistrust of the health care system on personal health practices and health outcomes in a prospective cohort of veterans with Type 2 Diabetes

DETAILED DESCRIPTION:
Background/Significance: Diabetes mellitus is a chronic and progressive disease that causes significant morbidity and mortality and increases health care utilization and costs in both Veteran Administration (VA) and non-VA settings. 1. Diabetes and its complications are more prevalent in minority populations. Black Americans have two-fold increased age adjusted rates of diabetes, are more likely to develop and experience greater disability from diabetes complications compared to White Americans. 1. Black Americans with diabetes have higher rates of retinopathy, end-stage renal disease, lower limb amputations, and overall death rates. 2. Therefore, diabetes is a significant public health problem and Black American patients have disproportionately higher morbidity and mortality than their White American counterparts.

Several factors have been postulated to explain the disproportionately higher morbidity and mortality from diabetes in Black Americans and these include their mistrust of the health care system. 3. It is thought that distrustful patients are less likely to seek routine medical care, take prescribed medications consistently, adhere to treatments recommendations, and maintain continuity with health care providers and health care systems. 4. Recent studies show that Black Americans are less trusting of physicians and the health care system. 5. However, little is known about the association between trust and diabetes outcomes and whether distrust of physicians and the health care system contributes to the observed racial/ethnic differences in diabetes outcomes.

Theoretical Framework: The conceptual and theoretical framework of this study is the revised behavioral model of health services use (Andersen 1974, 1968, 1983, 1995). The model posits that people's use of health services is a function of their predisposition to use services, factors that enable or impede use, and their need for care (Andersen 1995). Trust in physicians and the health system falls under health beliefs (attitudes toward health services), which is one of the predisposing factors that is thought to predict health services utilization and health outcomes. Thus, people with high levels of trust in physicians and the health care system are expected to have more effective access, appropriate health utilization, and better health outcomes. The model has been revised to include veteran-specific variables such as level of service entitlement, period of service, duration in the VA system, and disability status and to measure both health services use and health outcomes.

Research Design and Methods: This is a prospective cohort study with five hypotheses organized under their specific aims as follows:

Specific Aim #1: Determine racial/ethnic differences in trust in physicians and mistrust of the health care system among veterans with Type 2 Diabetes.

Hypothesis #1: There is a difference in mean scores on the general trust in physician scale (GTIPS) between White and Black American veterans with Type 2 diabetes.

Hypothesis #2: There is a difference in mean scores on the Health Care System Distrust Scale between White and Black American veterans with Type 2 diabetes.

Specific Aim #2: Determine the predictive power of trust in physicians and mistrust of the health care system on personal health practices and health outcomes in a prospective cohort of veterans with Type 2 Diabetes

Hypothesis #1: Controlling for predisposing, enabling, need, and veteran-specific factors, diabetic veterans with lower trust scores or higher mistrust scores will be less likely to keep office appointments, take prescribed medications, and adhere to diabetes self-management recommendations after 12 months of follow-up.

Hypothesis #2: Controlling for predisposing, enabling, need, and veteran-specific factors, diabetic veterans with lower trust scores or higher mistrust scores will have higher mean hemoglobin A1C, blood pressure, and LDL cholesterol levels after 12 months of follow-up.

Hypothesis #3: Controlling for predisposing, enabling, need, and veteran-specific factors, diabetic veterans with lower trust scores or higher mistrust scores will be less likely to accept influenza vaccination after 12 months of follow-up.

Study site & Subjects: Patients will be recruited from the Charleston VAMC. Equal number of White and Black American veterans aged 18 years and older with Type 2 Diabetes will be recruited. Race/ethnicity will be based on self-report. The diagnosis of type 2 Diabetes as well as health utilization and diabetes-specific health outcomes will be obtained from the VA electronic medical records system (CPRS). There are approximately 6,961 patients with Type 2 Diabetes at this site, of which 49.1% (3,417) are White Americans, 31.5% (2,189) are Black Americans, and 19.4% (1,355) are Hispanic or other. Approximately 97.5% are men and 90% are aged 50 years or older.

Sample size calculation:

Specific Aim #1: Sample Power V2.0 (SPSS) was used for sample size calculation based on the convention outlined by Cohen6. Overall experiment wise error was held to ?=0.05, and power to 80% using medium (0.25) effect sizes. Correction for multiplicity of tests (2 tests for primary hypotheses) involved using ?=0.025 (0.05/2). This yielded 125 patients per group. In addition, the sample was inflated to account for an estimated 20% attrition at 1 year of follow-up (death, relocation, or loss to follow-up). No more than 150 eligible patients need to be enrolled per group. Thus, 300 patients (150 Whites and 150 African Americans) will be recruited.

Specific Aim #2: The sample size determination for a reliable regression equation offered by Stevens7 is 15 subjects per predictor variable. Using this standard, a sample size of 300, as determined above, would allow the inclusion of 20 predictor variables. Because none of the hypotheses for Specific Aim 2 exceed 20 predictor variables, a sample of 300 will be adequate.

Survey Instruments: The GTIPS4 is a valid and reliable 11-item measure of general trust in physicians and the Health Care System Distrust Scale is a valid and reliable 10-item measure of mistrust of the health care system. Both instruments have been validated in Black and White Americans.

Statistical Analysis Plan: Descriptive statistics will be used to describe the characteristics of participants in the study.

Specific Aim #1: Mean scores on the trust and mistrust scales at baseline will be compared between White and Black Americans with the two-sample t-test and similar comparisons will be made while controlling for covariates (predisposing, enabling, need, and veteran-specific factors) using Analysis of Covariance (ANCOVA).

Specific Aim #2: Multiple linear regression will be used to test the effect of mean trust/mistrust scores on health utilization and mean hemoglobin A1C, blood pressure, and LDL cholesterol after 12 months of follow-up controlling for covariates. Similarly, multiple logistic regression will be used to test the effect of trust/mistrust on acceptance of the influenza vaccine controlling for covariates. STATA V8.0 will be used for data analysis and all tests will be two-tailed with overall p=0.05 for each hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Patients for this study will be recruited from the Ralph H. Johnson VAMC in Charleston, South Carolina.
* American veterans aged 18 years and older with Type 2 Diabetes will be recruited.

Exclusion Criteria:

* Children will not be included as this study pertains to type 2 diabetes, which is not a disease of children.
* Non-English speaking patients are excluded to eliminate bias in the response to questionnaires because these questionnaires have only been validated in English speaking patients.
* We decided to exclude cognitively impaired individuals because of the complexity of the survey instruments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: equal number of White and Black Americans over the age of 18 with Type II diabetes
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2004-11; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard E. Egede, MD MS, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the Charleston VAMC. Veterans with Type 2 Diabetes identified through the VA electronic medical resources system (CPRS) were consented and enrolled between November 2004 and February 2006.
Groups:
- White American Veterans: White American adult Veterans (age 18 or older) with type 2 diabetes
- Black American Veterans: Black American adult Veterans (age 18 or older) with type 2 diabetes
Period: Overall Study
Arm/Group | White American Veterans | Black American Veterans
Started | 150 | 150
Completed | 150 | 150
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants were adults (age 18 or older) with type 2 diabetes. All participants completed questionnaire, however, discrepancies in number of participants analyzed for specific measures is due to some participants choosing not to answer all questions. All participants are included in baseline measure for age.
Groups:
- Total: Total of all reporting groups
Arm/Group | White American Veterans | Black American Veterans | Total
Number analyzed (Participants) | 150 | 150 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.11 (9.49) | 63.78 (10.84) | 65.93 (10.41)
Gender [Number; unit: participants] — Discrepancies in number of participants analyzed is due to some participants choosing not to answer all questions.
  participants
    Female | 2 | 4 | 6
    Male | 143 | 142 | 285
Marital Status [Number; unit: participants] — Discrepancies in number of participants analyzed is due to some participants choosing not to answer all questions.
  participants
    Married | 101 | 84 | 185
    Not Married | 44 | 64 | 108
Diabetes Duration [Mean (Standard Deviation); unit: years] | 11.6 (11.1) | 10.0 (8.0) | 10.8 (9.7)
Education [Mean (Standard Deviation); unit: years] | 13.4 (2.9) | 12.3 (3.2) | 12.8 (3.1)
Work Status [Number; unit: participants] — Discrepancies in number of participants analyzed is due to some participants choosing not to answer all questions.
  participants
    Working | 39 | 34 | 73
    Retired | 71 | 50 | 121
    Disabled | 29 | 48 | 77
    Other | 4 | 7 | 11
Income [Number; unit: participants] — Discrepancies in number of participants analyzed is due to some participants choosing not to answer all questions.
  participants
    < $20,000 | 46 | 73 | 119
    $20,000-$34,999 | 49 | 32 | 81
    $35,000-$49,999 | 20 | 18 | 38
    $50,000-$74,999 | 14 | 13 | 27
    > $75,000 | 12 | 1 | 13
Comorbidity Index [Mean (Standard Deviation); unit: units on a scale] — Charlson Comorbidity Index is a valid and reliable weighted index that estimates the risk of death from comorbid disease. The 17-item questionnaire takes into account the number and the seriousness of various comorbid diseases. The total score ranges from 0-37 with higher scores indicating higher predicted mortality.
  units on a scale | 1.8 (1.3) | 2.0 (2.4) | 1.9 (1.9)

OUTCOME MEASURES:

1. Primary Outcome: General Trust in Physicians Scale (GTIPS)
Description: The GTIPS is a valid and reliable 11-item measure of general trust in physicians in the domains of dependability, confidence, and confidentiality of information. All items are fashioned in a 5-point Likert format with a minimum score of 11 and maximum of 55. Higher scores indicate more trust in physicians.
Time Frame: 12 months following enrollment
Population: Discrepancies in number of participants analyzed is due to some participants choosing not to answer all questions.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | White American Veterans | Black American Veterans
Number analyzed (Participants) | 144 | 145
units on a scale | 39.0 (9.7) | 39.5 (7.6)
Statistical Analysis 1: Comparison: White American Veterans vs Black American Veterans; Test type: Superiority or Other; p = 0.648, ANOVA

2. Secondary Outcome: Hemoglobin A1c
Time Frame: 12 months after enrollment
Population: Discrepancies in number of participants analyzed is due to some participants having no data in their medical record for this measure.
Measure: Mean (Standard Deviation); unit: % HbA1c
Arm/Group | White American Veterans | Black American Veterans
Number analyzed (Participants) | 141 | 146
% HbA1c | 6.8 (1.2) | 7.1 (1.4)
Statistical Analysis 1: Comparison: White American Veterans vs Black American Veterans; Test type: Superiority or Other; p = 0.14, ANOVA

3. Primary Outcome: Health Care System Distrust Scale
Description: Health Care System Distrust Scale is a valid and reliable 10-item measure of distrust of the health care system, measuring honesty confidentiality and confidence. All questions are measured on a Likert scale, with scores ranging from a minimum of 10 to a maximum of 50. Higher scores indicate more distrust in the health care system.
Time Frame: 12 months after enrollment
Population: Discrepancies in number of participants analyzed is due to some participants choosing not to answer all questions.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Black American Veterans: White American adult Veterans (age 18 or older) with type 2 diabetes
Arm/Group | White American Veterans | Black American Veterans
Number analyzed (Participants) | 143 | 144
units on a scale | 26.6 (7.4) | 26.3 (7.1)
Statistical Analysis 1: Comparison: White American Veterans vs Black American Veterans; Test type: Superiority or Other; p = 0.675, ANOVA

4. Secondary Outcome: Systolic Blood Pressure
Time Frame: 12-months after enrollment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | White American Veterans | Black American Veterans
Number analyzed (Participants) | 141 | 146
mmHg | 131.9 (14.6) | 135.7 (14.6)
Statistical Analysis 1: Comparison: White American Veterans vs Black American Veterans; Test type: Superiority or Other; p = 0.03, ANOVA

5. Secondary Outcome: Diastolic Blood Pressure
Time Frame: 12-months after enrollment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | White American Veterans | Black American Veterans
Number analyzed (Participants) | 141 | 146
mmHg | 71.1 (8.9) | 75.9 (8.8)
Statistical Analysis 1: Comparison: White American Veterans vs Black American Veterans; Test type: Superiority or Other; p < 0.001, ANOVA

6. Secondary Outcome: LDL-cholesterol
Time Frame: 12-months after enrollment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | White American Veterans | Black American Veterans
Number analyzed (Participants) | 138 | 146
mg/dL | 86.4 (22.5) | 101.2 (27.5)
Statistical Analysis 1: Comparison: White American Veterans vs Black American Veterans; Test type: Superiority or Other; p < 0.001, ANOVA

ADVERSE EVENTS:
Time Frame: time period of the study - 12-months
Arm/Group | White American Veterans | Black American Veterans
Serious Adverse Events (participants affected / at risk) | 0/150 | 0/150
Other Adverse Events (participants affected / at risk) | 0/150 | 0/150

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes